CLINICAL TRIAL: NCT00637065
Title: Use of the Endothelin-1 Antagonist Bosentan in Patients With Established Pulmonary Hypertension and Fibrotic Lung Disease. - A Randomised, Placebo-Controlled, Double-Blinded Study.
Brief Title: Bosentan in Pulmonary Hypertension in Interstitial Lung Disease Treatment Study
Acronym: B-PHIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Actelion (Industry)
Responsible Party: Royal Brompton Hospital NHS Trust, Royal Brompton Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007OE002B; REC number: 07/H0714/125; EudraCT no: 2007-001643-21
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis; Nonspecific Interstitial Pneumonia
Keywords: Pulmonary hypertension; Interstitial lung disease; Idiopathic pulmonary fibrosis; Nonspecific interstitial pneumonia; Bosentan; Endothelin receptor antagonists; Pulmonary vascular resistance
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Bosentan tablets (62.5mg bd for first 4 weeks, then 125mg bd as tolerated)
  Interventions: Drug: Bosentan
- 2 (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — Bosentan tablets - 62.5mg bd for first 4 weeks, then 125mg bd if tolerated until trial completion.
  Other Names: Tracleer
  Arms: 1
Drug: Placebo — Placebo tables - identical to active drug but without the active ingredient -
  Other Names: Placebo tablets
  Arms: 2

SUMMARY:
Over time, patients with fibrosing or interstitial lung disease (ILD) can develop high lung blood pressures (pulmonary hypertension), and this is associated with poorer prognosis and survival. It is thought that development of PH contributes to the deterioration and death of patients with ILD. Endothelin-1 (ET1) is a substance contributing to the development of both PH and ILD. Bosentan is a drug blocking the action of ET-1 by binding to its receptors. Bosentan clearly benefits patients with PH of unknown cause, or related to other diseases (such as heart conditions, or HIV) both alone and in combination with other treatments. In patients with fibrosing lung disease and PH, there have been no controlled treatment studies. Clearly it is important to evaluate the effectiveness of bosentan in these patients.

This study aims to determine the ability of bosentan to reduce high blood pressure in the lungs (pulmonary hypertension) in patients with scarring (fibrosing) lung disease. It is a placebo-controlled double blinded study for 16 weeks (and it is proposed to follow patients in a 16 week open-label phase with bosentan therapy).

DETAILED DESCRIPTION:
• Purpose: High blood pressure in the lungs or pulmonary hypertension (PH) is a common complication of fibrosing (or interstitial, ILD) lung disease. When present, it is associated with markedly reduced prognosis and survival. Endothelin-1 (ET-1)is over-expressed in patients with PH and ILD, and is thought to play a role in the development of both conditions. Bosentan blocks the action of ET-1, and has been shown to be beneficial in patients with PH from an unknown cause, or related to other conditions (such as heart conditions, connective-tissue disease, and HIV). It is important to establish whether bosentan treatment also benefits patients with PH and ILD.

This study addresses the effectiveness of bosentan in the context of PH and ILD.

• Objective: To examine the ability of bosentan to reduce high blood pressure in the lungs in patients with fibrosing lung diseases and pulmonary hypertension.

• Design: This is a multi-centre, randomised, double-blinded, placebo-controlled study looking at the effect of bosentan in patients with fibrotic lung disease and PH.

• Methodology: Patients will be recruited from outpatient ILD and PH clinical services and will be consented prior to entering the study. We propose to study 48 patients over a 16 week period. Patients will be included in the study if they have fibrosing lung disease (specifically: idiopathic pulmonary fibrosis or idiopathic fibrosing non-specific pneumonitis) and have PH as determined by measurement on right heart catheter (mean pulmonary artery pressure >=25mmHg, pulmonary capillary wedge pressure =<15mmHg).

Patients will enter a 2 week screening period during which they will have a full medical history and examination. If they have not already had clinically important investigations ( echocardiogram, cardiac MRI, overnight oximetry) within the previous 6 weeks and CT scan within the last 3 months, these will be performed.

The patient will have a baseline 6 minute walk test, ECG (heart tracing), blood tests and pulmonary blood flow study (breath test) and lung function tests (breathing tests) and complete a quality of life questionnaire. The patient will then be randomised to bosentan or placebo (2:1)at the baseline visit. Patients will be followed every 4 weeks with physical examination, and blood tests.

At week 16, the initial investigations (including right heart catheter, lung function, pulmonary blood flow, 6-minute walk, blood tests, echocardiogram and cardiac MRI and complete a quality of life questionnaire) will be repeated.

Patients will be offered treatment with open-labelled bosentan therapy until the results of the trial become available up to a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >=18yrs, <80yrs
2. Patients with idiopathic pulmonary fibrosis (IPF) or idiopathic fibrotic non-specific interstitial pneumonitis (NSIP) confirmed by their respiratory physician according to ATS/ERS criteria.
3. Patients with pulmonary hypertension on right heart catheter (mean pulmonary arterial pressure >=25mmHg with pulmonary artery occlusion pressure, left atrial pressure or left ventricular end-diastolic pressure <15mmHg).
4. Patients providing written informed consent.

Exclusion Criteria:

1. Patients <18, >80yrs.
2. Patients with unstable disease, or an acute exacerbation of their underlying fibrotic lung disease.
3. Patients with significant other organ co-morbidity including hepatic or renal impairment.
4. Patients with systolic BP < 85mmHg
5. Patients with other conditions that may affect the ability to perform a 6-minute walk test.
6. Patients unable to provide informed consent and comply with the patient protocol.
7. Patients receiving excluded medications (including: epoprostenol, or prostacyclin analogues, phosphodiesterase inhibitors, other endothelin receptor antagonists, drugs with potential interaction with bosentan such as glibenclamide, fluconazole, cyclosporin A, or tacrolimus, and other investigational agents).
8. Patients with planned surgical intervention during the study period.
9. Pregnant patients or women of child-bearing age, who are not using a reliable contraceptive method.
10. Patients with clinically overt ischaemic heart disease.
11. Patients with predominant emphysema on high resolution CT scan (emphysema greater in extent than interstitial changes).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is a fall in pulmonary vascular resistance (PVR) of 20% over 16 weeks. | 16 weeks

SECONDARY OUTCOMES:
mean Pulmonary arterial Pressure | 16 weeks
Six minute walk distance | 16 weeks
Quality of life scores (Camphor questionnaire) | 16 weeks
Pulmonary function (DLco, FVC and PaO2) | 16 weeks
Pulmonary blood flow | 16 weeks
Right ventricular mass (Cardiac MRI) | 16 weeks
BNP | 16 weeks
Progression free survival | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Wort, FRCP PhD, Principal Investigator — Royal Brompton Hospital, London; Athol U Wells, MD FRCP FRCR, Principal Investigator — Royal Brompton Hospital, London; Luke Howard, DPhil MRCP, Principal Investigator — Hammersmith Hospitals NHS Trust; Brendan Madden, MD MSc FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - St George's Hospital, London, London
  - Royal Brompton Hospital, London, London
  - Hammersmith Hospital, London, London

REFERENCES:
- [Derived] Corte TJ, Keir GJ, Dimopoulos K, Howard L, Corris PA, Parfitt L, Foley C, Yanez-Lopez M, Babalis D, Marino P, Maher TM, Renzoni EA, Spencer L, Elliot CA, Birring SS, O'Reilly K, Gatzoulis MA, Wells AU, Wort SJ; BPHIT Study Group. Bosentan in pulmonary hypertension associated with fibrotic idiopathic interstitial pneumonia. Am J Respir Crit Care Med. 2014 Jul 15;190(2):208-17. doi: 10.1164/rccm.201403-0446OC. PMID 24937643